CLINICAL TRIAL: NCT02252822
Title: Does Offering Adolescents Anonymous Access to Online CBT Self-Help for Bulimia Nervosa Improve Engagement in Treatment-Pilot Study
Brief Title: Improving Treatment Engagement for Adolescents With Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Psychiatrist, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59093006
Record Dates: First submitted 2014-06-26; First posted 2014-09-30 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Self Help; Anonymous CBT
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Overcoming Bulimia Online Programme (Experimental): This treatment incorporates a combination of cognitive-behavioral, motivational and education strategies. The program will be presented in 8 collaborative, multi-media, web based CBT sessions for BN.
  Interventions: Behavioral: Overcoming Bulimia Online Programme

INTERVENTIONS:
Behavioral: Overcoming Bulimia Online Programme

SUMMARY:
Although 4.7% of adolescents suffer from symptoms of bulimia nervosa (BN), only 1/5 seek treatment. Hesitation to seek treatment is likely related to ego-syntonicity and fear of disclosing symptoms to parents and clinicians. Furthermore, the physical symptoms of BN often go unnoticed by parents and clinicians.

In order to eliminate the barriers that prevent adolescents from seeking treatment, this study will offer anonymous access to online self-help cognitive behavioral therapy (CBT) for BN. Online CBT (traditional, non-anonymous delivery) has been found to be effective and acceptable treatment for adolescents with BN. Furthermore, in adults, this method has been found to be as effective as specialized treatments, and more cost efficient.

To remain anonymous and accessible, the self-help approach in this study will be provided in a non-guided, or pure format (only online sessions). Studies support that a pure self-help methodology is as effective as a guided version.

Although anonymity may improve accessibility, this study design could also pose challenges in areas such as recruitment, treatment completion and obtaining adequate informed consent. Therefore, before embarking on a larger randomized control trail, we would like to propose a small, non-controlled feasibility study to assess potential issues in these areas.

Primary hypotheses:

Recruitment: Based on communication with public health nurses in the high schools we plan to recruit from, we hypothesize that it is feasible to recruit 1-5 adolescents over a 4-month period from each of the 5 schools, and 1-5 from social media outlets such as Instagram, Twitter, Facebook for a total of 5 participants over a 4-month period.

Treatment completion: Based on pervious studies of self-help for adolescent bulimia, we hypothesize that approximately 15% of participants will not complete any sessions, and many will only complete about half of the sessions.

Informed consent: Based on information from large randomized control studies in the UK, we hypothesize that adolescents will be capable of providing online consent, and that we will be able to adequately obtain consent without verbally communicating with participants.

Secondary hypothesis:

We hypothesize a non-guided (pure) version of online CBT-BN offered in an anonymous manner will decrease BN symptoms after treatment completion, and at 3-month follow-up compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with symptoms of BN (full threshold or subthreshold) defined by self-reported symptoms of binging and compensatory behaviours (self-induced vomiting, laxative abuse, diet pills, and diuretics). Excessive exercise and fasting will not be included due to the potential for subjectively in a self-report format.
* Ages of 16-18.
* Consent from the adolescent.

Exclusion Criteria:

* Adolescent is actively engaged in psychological treatment for bulimia nervosa.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Recruitment | 4 months
  The rate of recruitment per month will be compared to standard research recruitment rates, and extrapolation of these data will be a means of assessing feasibility for recruitment for a larger RCT.
Treatment completion | 2 months
  The medium number of completed online sessions will be compared to previous studies on self-help online CBT for BN in order to ensure at least comparable completion rates are achieved using our novel treatment design. Participants will be provided with a feedback form following treatment completion in order to assess treatment satisfaction and adherence.
Informed consent | Baseline
  The informed consent process will be evaluated based on the participants ability to effectively answer online questions aimed at determining an understanding of the consent process. Participants would need to answer all questions correctly in order to be deemed capable of consenting.

SECONDARY OUTCOMES:
Eating Disorder Examination-Questionnaire Version (EDE-Q) | Baseline, 8weeks (post-intervention), 3-month follow-up
  This measure will asses effectiveness of online self-help CBT-BN in improving BN symptoms. The EDE-Q measures 4 areas of eating disorder pathology (eating concern, weight concern, dietary restraint and shape concern).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Keshen, MD, FRCPC, Principal Investigator — Capital Health, Canada
Locations (1):
- Capital Health District Health Authority, Halifax, Nova Scotia, Canada